CLINICAL TRIAL: NCT03780049
Title: Hepatic Artery Infusion Chemotherapy Plus Recombinant Human Type-5 Adenovirus vs Hepatic Artery Infusion Chemotherapy Alone for Unresectable Hepatocellular Carcinoma at Barcelona Clinic Liver Cancer A-B Stage
Brief Title: HAIC Plus H101 vs HAIC Alone for Unresectable HCC at BCLC A-B
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCC-S032
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic artery infusion chemotherapy; Oxaliplatin, 5-fluorouracil and leucovorin; Recombinant Human Type-5 Adenovirus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil; Leucovorin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC plus H101 (Experimental): Patients receive oxaliplatin, 5-fluorouracil and leucovorin and recombinant human type-5 adenovirus 0.5ml via hepatic artery
  Interventions: Procedure: HAIC of FOLFOX; Drug: H101
- HAIC (Active Comparator): Patients receive oxaliplatin, 5-fluorouracil and leucovorin and normal saline via hepatic artery
  Interventions: Procedure: HAIC of FOLFOX; Drug: Placebos

INTERVENTIONS:
Procedure: HAIC of FOLFOX — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Other Names: Hepatic artery infusion chemotherapy of oxaliplatin , fluorouracil, and leucovorin
Drug: H101 — Patients receive H101 0.5ml dissolved in 10ml normal saline in each session of HAIC
  Other Names: Recombinant Human Type-5 Adenovirus
  Arms: HAIC plus H101
Drug: Placebos — Patients receive normal saline 10ml in each session of HAIC
  Other Names: normal saline
  Arms: HAIC

SUMMARY:
Hepatic artery infusion chemotherapy (HAIC) is effective and safe for hepatocellular carcinoma (HCC). Recombinant Human Type-5 Adenovirus (H101) is safe for HCC. The purpose of this study is to evaluate the efficacy and safety of HAIC combined with H101 compared with HAIC alone in patients with unresectable hepatocellular carcinoma (HCC) at barcelona clinic liver cancer A-B stage.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* Single lesion with tumor size larger 7cm or multiple lesions
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* BCLC A-B stage
* The following laboratory parameters:

Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Patients complicated by history of heart disease, history of gastrointestinal bleeding within 1 month, severe infection (> grade 2 National Cancer Institute [NCI] -common Terminology Criteria for Adverse Events [CTCAE] version 4.0) or other serious associated diseases will not be able to tolerate treatment
* With other malignant tumors
* Known or suspected allergy to the investigational agents or any agent given in association with this trial
* History of organ allograft
* Pregnant or lactating woman
* patients with poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Number of adverse events | 30 days
  Postoperative adverse events were graded based on CTCAE v4.03
Conversion rate to resection | 24 months
  Patients receive subsequent resection.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China